CLINICAL TRIAL: NCT00461968
Title: Genetic Determinanats of Cardiovascular Risk Factors: Comparison of Efficacy and Safety of Ezetimibe or Statin Monotherapy to Co-Administration of Both
Brief Title: Comparison of Efficacy and Safety of Ezetimibe or Statin Monotherapy to Co-Administration of Both
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Donald W. Reynolds Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 072004-28
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Cholesterol, LDL
Keywords: Cholesterol; LDL; Ezetimibe; Statin; Zetia; Zocor; Simvastin
MeSH Terms: interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Ezetimibe and Simvastatin

SUMMARY:
The purpose of this study is to compare the percent change in LDL cholesterol induced by ezetimibe or simvastatin monotherapy and by co-administration of both agents in Black, White and Hispanic men. Ezetimibe is a drug that blocks sterol absorption and simvastatin blocks hepatic cholesterol biosynthesis. The hypothesis to be tested is that Blacks are likely to be more responsive to LDL lowering by ezetimibe than statins because Blacks have a low production of cholesterol.

DETAILED DESCRIPTION:
Statins effectively lower plasma LDL cholesterol levels at the lowest recommended doses, and subsequent doubling of the dosage results in a modest additional reduction of about ~6%. A large inter-individual variability in the magnitude of the LDL-lowering response is seen in patients taking statins, as revealed by data provided to the P.I. by Merck & Co. Inc. Mean reductions in plasma levels of LDL-C and the variation in response (SD) are provided for ~300 subjects taking only simvastatin, only ezetimibe or both ezetimibe and simvastatin. The mechanisms responsible for this inter-individual variability in lipid-lowering response is not known. The effect of ethnicity on the statin-associated LDL-lowering has only been examined in one study. In this study, directed attempts were made to implement the NCEP guidelines for secondary prevention using statins. Fewer Blacks than Whites reached the goal of treatment for plasma LDL-C levels, despite being seen more frequently in the clinic and having their lipoproteins measured more often. It was proposed that this difference was due to lower compliance with the drug regimen among Blacks. An alternative explanation for the ethnic difference in response to therapy is that the effectiveness of statins differs between ethnic groups.

We hypothesize that Blacks are likely to be more responsive to agents that inhibit cholesterol absorption and less responsive to agents that interfere with cholesterol synthesis. This hypothesis is also based on the results of a recent study conducted in our laboratory that showed lower levels of lathosterol in Blacks than in Whites. Lathosterol is a precursor of cholesterol and therefore it is a marker of de novo synthesis of the sterol. In contrast, campesterol is a plant sterol and its plasma levels are assumed to be indicators of sterol absorption. To directly address the study question, an intervention study that compares the relative efficacy of ezetimibe and simvastatin will be carried out. In this aim we will answer the following questions:

* Do Blacks, Whites and Hispanics respond differently to simvastatin and ezetimibe?
* Do baseline levels of noncholesterol sterols and/or the campesterol:lathosterol ratios predict responsiveness to cholesterol-lowering drugs?
* Does the low level of plasma lathosterol in Blacks reflect reduced rates of cholesterol synthesis secondary to increased cholesterol absorption, and is the relative responsiveness to the two different classes of LDL-lowering agents used in the clinical trial related to the balance between cholesterol absorption and synthesis in an individual?

The ultimate goal is to identify genetic or metabolic indices that can be used to individualize cholesterol lowering therapy, allowing the most effective therapeutic regimen to be selected. This is particularly important if long-term lipid lowering therapy is to be used in individuals whose short-term cardiovascular risk is low since it would be particularly desirable to use the most effective drugs at the lowest doses in this setting.

This will be a randomized, double-blind, placebo-controlled, 4-period, crossover study of 26 weeks duration comprising a 3-day screening period; a 2-week, single-blind placebo run-in period; and four 6-week, double-blind treatment periods. Each individual will be randomized to one of the four treatment sequences. Randomization will be stratified by race (Black/White); both Black and White subjects will be allocated in a 1:1:1:1 ratio to the 4 treatment sequences. The Allocation schedule will be generated at Merck and Merck will maintain the blinding. There are 10 required clinic visits (visit 1,2,4,5,7,8,10,11,13,14), and 5 telephone contacts (visit 3,6,9,12) at the mid-point of each treatment period to review compliance with diet, study medications, and alcohol consumption requirements. A post-study follow-up will also be conducted via telephone for serious adverse experience review (visit 15). Total visits will be 15 (10 clinic and 5 telephone) Each treatment period will last about 6 weeks. During the screening visit, subjects will undergo a physical exam, dietary assessment, vital signs (blood pressure, heart rate, and respirations), and provide blood (3 tablespoons) sample for routine chemistries (metabolic comprehensive panel), complete blood count, liver function tests, thyroid test, and plasma cholesterol, triglyceride and lipoprotein cholesterol measurement by beta-estimation) levels, and a urine sample. Subjects meeting eligibility criteria will be scheduled to return for Visit 2 to begin a two-week single-blind placebo run-in phase. At Visit 3, subjects who, by pill count, miss no more than two tablets of the single-blind study medication will be randomized to one of the 4 treatment sequences. Subjects will take 2 pills each day. Vital signs will be performed at each visit. A physical will be completed at the end of the study. Serum chemistry measurements, plasma cholesterol and triglyceride levels, lipoprotein cholesterol by beta-quantitation, measurement of apolipoprotein B and measurement of non-cholesterol sterols will be measured at all visits (3-4 tablespoons of blood will be drawn). The analyses will be repeated in a separate plasma sample if the data are inconsistent or needs verification. Circulating levels of noncholesterol sterols will be measured by gas chromatography and mass-spectrometry, a routine procedure in our laboratory, in the same samples. Investigators will be blinded to lipid/lipoprotein values after Visit 1. Hematology and urinalysis will be performed at Visits 1 and 14. Dietary counseling will be provided during the study. Also, DNA will be extracted from blood samples obtained during the trial to examine genes that control cholesterol metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Black, white and hispanic males between the ages of 20 to 70 years
* In good general health
* Having a body mass index (BMI) between 20 and 35 kg/m2
* Plasma LDL-C concentrations greater than or equal to 130 mg/dl but less than or equal to 175 mg/dL
* TG (triglyceride) levels less than or equal to 250 mg/dL.

Exclusion Criteria:

* Any condition that would be likely to render the individual unable to complete the study
* Hypersensitivity to HMG-CoA reductase inhibitors
* Poor mental function, drug or substance abuse, or unstable psychiatric illnesses that may interfere with optimal participation in the study
* Treatment with another investigational drug within 30 days prior to Visit 1
* Alcohol consumption >14 drinks per week
* Phytosterol/phytostanol-containing products including margarines within 2 weeks
* History of CHD, peripheral vascular disease, cerebrovascular disease, CHF, or uncontrolled arrhythmias
* Creatinine >1.5 mg/dL, nephrotic syndrome, or other renal disease
* Fasting plasma glucose (FPG) >126 mg/dL or history of diabetes
* Abnormal TSH
* Uncontrolled hypertension (systolic BP >160 mm Hg and/or diastolic BP >100 mm Hg)
* Known active liver diseases or elevated serum transaminases (ALT and AST >1.5 times the upper limit of normal)
* Digestive disorders or any abdominal surgery within the past 6 months
* Cancer within the past 5 years (except for skin cancer)
* HIV, HBV, or HCV positive
* Lipid-lowering agents: bile-acid binding resins, HMG-CoA reductase inhibitors, ezetimibe, niacin (>200 mg/day), cholestin, fish oil, and fibrates, or cholesterol absorption inhibitors (e.g., neomycin) taken within 8 weeks prior to Visit 1
* Medications that are potent inhibitors of CYP3A4 (cyclosporine, systemic itraconazole or ketoconazole, erythromycin or clarithromycin, nefazodone, verapamil, amiodarone, and protease inhibitors)
* Anti-obesity medications: orlistat or sibutramine taken within 8 weeks prior to Visit 1
* Systemic corticosteroids.

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoints of the study will be the percent change in plasma LDL-C concentrations in response to each agent.
The treatment effect for each individual will be the percent reduction achieved with each agent.

CONTACTS AND LOCATIONS:
Overall Officials: Helen H Hobbs, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States